CLINICAL TRIAL: NCT04718402
Title: A Multicenter, Open-label, Single-arm, Phase Ib Study to Evaluate the Safety and Efficacy of Mitoxantrone Hydrochloride Liposome Injection in Subjects With Advanced Gastric Carcinoma
Brief Title: A Study of Mitoxantrone Hydrochloride Liposome Injection in the Treatment of Advanced Gastric Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor has adjusted its R&D strategy.
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE071-CSP-014
Record Dates: First submitted 2020-12-14; First posted 2021-01-22 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2021-05

CONDITIONS: Advanced Gastric Carcinoma
MeSH Terms: interventions — Injections, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitoxantrone Hydrochloride Liposome Injection (Experimental): Subjects with advanced gastric carcinoma will receive 20mg/m2Mitoxantrone Hydrochloride Liposome every 21 days (a cycle) for a maximum of 8 cycles.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome, intravenous injection

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome, intravenous injection — All subjects will receive Mitoxantrone Hydrochloride Liposome 20 mg/m2, IV, on day 1 of each 21-day cycle (q3w).

SUMMARY:
This is a multicenter, open-label, single-arm, phase Ib study to evaluate the safety and efficacy of Mitoxantrone Hydrochloride Liposome in subjects with advanced gastric carcinoma.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm, phase Ib study to evaluate the safety and efficacy of Mitoxantrone Hydrochloride Liposome in subjects with advanced gastric carcinoma. At least 30 subjects will be recruited in this study. The subjects will receive Mitoxantrone Hydrochloride Liposome 20 mg/m2 by an intravenous infusion (IV), every 21 days (q3w, 1 cycle). All patients will receive the treatment until disease progression, intolerable toxic reaction, death, or withdrawal by investigator or patient decision (a maximum of 8 cycles).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent;
2. Age ≥18, without gender limitation;
3. Histologically confirmed diagnosis of unresectable locally advanced or metastatic gastric carcinoma, including gastroesophageal junction carcinoma;
4. Suitable to receive the study drug as decided by the investigator;
5. At least one measurable lesion according to RECIST v1.1;
6. ECOG performance status of 0 to 2;
7. Life expectancy ≥ 12 weeks;
8. AEs from the previous treatment have resolved to ≤ Grade 1 based on CTCAE (except for the toxicity without safety risk judged by the investigator, such as hair loss, hyperpigmentation);
9. Adequate organ function;
10. Subjects of childbearing potential must agree to use effective contraceptive measures. Female subjects must have a negative pregnancy test before enrolment;
11. Fully comply with the protocol.

Exclusion Criteria:

1. History of allergy to mitoxantrone hydrochloride or any excipients of the study drug;
2. Untreated or symptomatic central nervous system (CNS) metastases;
3. Amenable to curative surgery ( radical excision);
4. Pleural effusion, pericardial effusion or peritoneal effusion with overt clinical symptoms (except for those have a drainage within 1 month before screening, asymptomatic and the effusion only detectable by imageological examination);
5. Intestinal obstruction with overt clinical symptom and requiring treatment;
6. CTCAE Grade 3 or Grade 4 gastrointestinal hemorrhage within 12 weeks prior to the first dose administration;
7. History of allotransplantation;
8. Known hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or other active viral infection;
9. Serious infection or interstitial pneumonia within 1 week prior to the first dose administration;
10. Use of other anticancer treatment within 4 weeks prior to the first dose administration;
11. Enrolled in any other clinical trails and had recieved treatment within 4 weeks prior to the first dose administration;
12. Major surgery within 3 months prior to the first dose administration, or have a surgical schedule during the study period;
13. Thrombosis or thromboembolism within 6 months prior to screening;
14. History of, or known additional malignant tumor within 3 years, except for tumors have been cured and have not recurred, and carcinoma in situ;
15. Impaired cardiac function or serious cardiac disease;
16. Previous treatment with adriamycin or other anthracyclines, and the total cumulative dose of prior adriamycin or equivalent is >350 mg/m2.
17. Pregnant or lactating female;
18. Serious and/or uncontrolled systemic diseases;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
adverse events (AEs) | From the initiation of the first dose to 28 days after the last dose, assessed up to 36 months
  The incidence and severity of AEs, abnormalities in physical exams, vital sign assessments, clinical laboratory assessments, ultrasonic cardiograms (UCGs) and electrocardiographs (ECGs).

SECONDARY OUTCOMES:
overall response rate (ORR) | From the enrollment to the final documentation of response of the last subject (assessed up to 36 months)
  To investigate the preliminary antitumor efficacy
duration of response (DoR) | From the enrollment to death, lost to follow-up, withdrawal, or study end, whichever occurred first, assessed up to 36 months
  To investigate the preliminary antitumor efficacy
duration of complete response (DCR) | From the enrollment to the final documentation of response of the last subject (assessed up to 36 months)
  To investigate the preliminary antitumor efficacy
progression-free survival (PFS) | From the enrollment to death, lost to follow-up, withdrawal, or study end, whichever occurred first, assessed up to 36 months
  To investigate the preliminary antitumor efficacy
overall survival (OS) | From the enrollment to death, lost to follow-up, withdrawal, or study end, whichever occurred first, assessed up to 36 months
  To investigate the preliminary antitumor efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Jieer Ying, Doctor, Principal Investigator — Cancer Hospital of The University of Chinese Academy of Science
Locations (9):
- China (9):
  - Beijing Luhe Hospital Capital Medical University, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The Fourth Hospital of Hebei Medical University and Hebei Cancer Hospital, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Cancer Hospital of The University of Chinese Academy of Science, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang